CLINICAL TRIAL: NCT03267576
Title: Canagliflozin Continuous Glucose Monitoring (CANA CGM) Trial: A Pilot Randomized, Double-Blind, Controlled, Crossover Study on the Effects of the SGLT-2 Inhibitor Canagliflozin (vs. the DPP-4 Inhibitor Sitagliptin) on Glucose Variability in Mexican Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin
Brief Title: An Efficacy Study of Canagliflozin or Sitagliptin to Determine Glucose Variability in Mexican Participants With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin
Acronym: COMETA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR108346; 28431754DIA4026 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Results first posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive metformin monotherapy at stable doses (greater than or equal to [>=] 1500 milligram per day [mg/day]) orally once daily with canagliflozin 300 milligram (mg) tablet orally once daily (Treatment A) from Day 0 to 27 (treatment period 1), followed by sitagliptin 100 mg tablet orally once daily with metformin >=1500 mg/day (Treatment B) from Day 44 to 71 (treatment period 2), under fasted condition. A washout period of at least 16 days (from Days 28 to 43) of metformin monotherapy will be maintained between each treatment period.
  Interventions: Drug: Canagliflozin 300 mg; Drug: Sitagliptin 100 mg; Drug: Metformin
- Treatment Sequence BA (Experimental): Participants will receive treatment B from Day 0 to 27 (treatment Period 1), followed by treatment A from Day 44 to 71 (treatment period 2), under fasted condition. A washout period of at least 16 days (from days 28 to 43) of metformin monotherapy will be maintained between each treatment period.
  Interventions: Drug: Canagliflozin 300 mg; Drug: Sitagliptin 100 mg; Drug: Metformin

INTERVENTIONS:
Drug: Canagliflozin 300 mg — Participants will receive canagliflozin 300 mg oral tablet once-daily for 28 days.
  Other Names: JNJ-28431754
Drug: Sitagliptin 100 mg — Participants will receive sitagliptin 100 mg oral tablet once-daily for 28 days.
Drug: Metformin — Participants will receive metformin at a stable dose of >= 1500 mg/day throughout the study including the washout period between each intervention.

SUMMARY:
The main purpose of this study is to assess the effects of 4 weeks each of daily treatment with canagliflozin 300 milligram (mg) versus sitagliptin 100 mg as treatment adjuncts to metformin (at stable dosages) on intrapatient glycemic coefficient of variation (CV), expressed as a ratio percentage of standard deviation (SD) to mean glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Inadequate glucose control while using metformin monotherapy (MET) for at least 8 weeks at stable daily doses of at least 1500 milligram (mg) before screening visit (Visit 1)

  a. Hemoglobin A1c (HbA1c) equal to (=) 7.5 percent (%) to 10.5% at Visit 1
* Adequate qualifying continuous glucose monitoring (CGM) reading during the pre-randomization (selection) phase
* Estimated glomerular filtration rate (eGFR) of at least 60 milliliter/minute (mL/min)/1.73 meter square (m^2) at Visit 1
* Body mass index of 22 through 45 kilogram per meter square (kg/m^2) at Visit 1

Exclusion Criteria:

* History of any of the following (at Visit 1):

  1. Diabetic ketoacidosis (DKA)
  2. Type 1 diabetes mellitus (T1DM)
  3. Pancreatic (for example, Beta-islet cell) transplantation
  4. Diabetes secondary to pancreatitis or pancreatectomy
  5. Personal history of, or ongoing, pancreatitis
  6. One or more episodes of severe hypoglycemia (requiring assistance from others), as documented in the history obtained at Visit 1
  7. Hereditary glucose-galactose malabsorption or primary renal glucosuria
* Repeated fasting plasma glucose (FPG) or fasting self-monitored blood glucose (SMBG) greater than (>) 270 milligram per deciliter (mg/dL) during the pre-treatment phase
* Treatment with any other oral or parenteral antidiabetic medications different from metformin monotherapy, including but not limited to Dipeptidyl peptidase-4 (DPP-4) inhibitors, Sulphonylureas, thiazolidinediones, insulins and Glucagon-like peptide-1 receptor agonist (GLP-1RAs); Sodium-glucose co-transporter 2 (SGLT-2) inhibitors and investigational agents
* Received an investigational drug or vaccine or used an invasive investigational medical device within 30 days before the planned first dose of study drug
* Current use of "natural medicines" or natural medicinal products for diabetes (for example, cactus-derived nutrients, celery)

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- Mexico (5):
  - Consultorio Privado, Guadalajara
  - Investigación Clínica Especializada, Guadalajara
  - Consultorio Privado en Unidad de Patología Clínica, Guadalajara
  - Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán, Mexico City
  - Hospital Universitario 'Dr. Jose Eleuterio Gonzalez', Monterrey

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 64 participants were enrolled in this study but 1 participant has withdrawn consent before assigning to any study treatment hence, 63 participants were randomized to study treatment arms.
Groups:
- Treatment Sequence AB: Participants received metformin monotherapy at stable doses (greater than or equal to [>=] 1500 milligram per day [mg/day]) orally once daily with canagliflozin 300 milligram (mg) tablet orally once daily (Treatment A) from Day 0 to 27 (treatment period 1), followed by sitagliptin 100 mg tablet orally once daily with metformin >=1500 mg/day (Treatment B) from Day 44 to 71 (treatment period 2), under fasted condition with a washout period of at least 16 days (from Days 28 to 43) along with ongoing metformin monotherapy.
- Treatment Sequence BA: Participants received metformin monotherapy at stable doses >=1500 mg/day with sitagliptin 100 mg tablet orally once daily (Treatment B) from Day 0 to 27 (treatment Period 1), followed by metformin >= 1500 mg/day orally once daily with canagliflozin 300 mg tablet orally once daily (Treatment A) from Day 44 to 71 (treatment period 2), under fasted condition with a washout period of 16 days (from days 28 to 43) along with ongoing metformin monotherapy.
Period: Period 1: Day 0 to 27
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Started | 31 | 32
Completed | 31 | 32
Not Completed | 0 | 0
Period: Washout Period: 16 Days
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Started | 31 | 32
Completed | 31 | 32
Not Completed | 0 | 0
Period: Period 2: Day 44 to 71
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Started | 31 | 32
Completed | 30 | 30
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all participants who received at least one dose of medication and in whom CGM recordings at baseline and after each active treatment were successful (greater than [>] 70 percent (%) of tracings available).
Groups:
- Treatment Sequence AB: Participants received metformin monotherapy at stable doses (greater than or equal to [>=] 1500 milligram per day [mg/day]) orally once daily with canagliflozin 300 milligram (mg) tablet orally once daily (Treatment A) from Day 0 to 27 (treatment period 1), followed by sitagliptin 100 mg tablet orally once daily with metformin >=1500 mg/day (Treatment B) from Day 44 to 71 (treatment period 2), under fasted condition with a washout period of at 16 days (from Days 28 to 43) along with continued metformin monotherapy.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence AB | Treatment Sequence BA | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.03 (6.237) | 44.84 (9.088) | 45.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 17 | 18 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Mexican mestizo | 31 | 32 | 63
  Caucasian | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Afro-American | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: Meter] | 1.63 (0.10) | 1.64 (0.10) | 1.63 (0.10)
Weight [Mean (Standard Deviation); unit: Kilogram] | 84.01 (15.86) | 88.96 (14.17) | 86.52 (15.11)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycemic Coefficient of Variation (CV) in Treatment Period 1
Description: Continuous blood glucose monitoring was done in participants using continuous glucose monitoring (CGM) determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and after each active treatment. Glucose coefficient of variation (CV) was calculated based on CGM data dividing the standard deviation of blood glucose values by the mean of the corresponding glucose readings. The participants were analyzed according to treatment received in treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27)
Population: Intent-to-treat (ITT) analysis set included all participants who received at least one dose of medication and in whom CGM recordings at baseline and after each active treatment were successful (greater than [>] 70% of tracings available).
Measure: Mean (Standard Deviation); unit: Percentage of CV
Groups:
- Treatment Sequence AB: Participants received metformin monotherapy at stable doses (greater than or equal to [>=] 1500 milligram per day [mg/day]) orally once daily with canagliflozin 300 milligram (mg) tablet orally once daily (Treatment A) from Day 0 to 27 (treatment period 1), followed by sitagliptin 100 mg tablet orally once daily with metformin >=1500 mg/day (Treatment B) from Day 44 to 71 (treatment period 2), under fasted condition with a washout period of 16 days (from Days 28 to 43) along with ongoing metformin monotherapy.
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Percentage of CV | -0.69 (5.17) | 0.24 (10.23)

2. Primary Outcome: Change From Baseline in Glycemic Coefficient of Variation (CV) in Treatment Period 2
Description: Continuous blood glucose monitoring was done in participants using CGM determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and after each active treatment. Glucose coefficient of variation was calculated based on CGM data dividing the standard deviation of blood glucose values by the mean of the corresponding glucose readings. The participants were analyzed according to treatment received in treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 2 (Days 66 to 71)
Population: ITT analysis set included all participants who received at least one dose of medication and in whom CGM recordings at baseline and after each active treatment were successful (>70% of tracings available).
Measure: Mean (Standard Deviation); unit: Percentage of CV
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Percentage of CV | -1.26 (7.41) | 0.77 (6.16)

3. Secondary Outcome: Change From Baseline in Glycemic Standard Deviation (SD) for 24-hour Glucose Profile
Description: Glycemic standard deviation for 24-hour glucose profile (glycemic variability), as measured by CGM was determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants who received the study drug in the treatment period 1 and 2 as per the sequence were reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: Per-protocol (PP) analysis set included all ITT participants without a major protocol violation, where ITT population included all participants who received at least one dose of medication and in whom CGM recordings at baseline and after each active treatment were successful.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
mg/dL
  Treatment Period 1 | -7.64 (6.56) | -8.40 (11.07)
  Treatment Period 2 | -8.53 (10.35) | -7.13 (12.00)

4. Secondary Outcome: Change From Baseline in Mean 24-hour Glucose Profile
Description: Mean 24-hour glucose profiles as measured by CGM was determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 and treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: PP analysis set included all ITT participants without a major protocol violation, where ITT population included all participants who received at least one dose of medication and in whom CGM recordings at baseline and after each active treatment were successful.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
mg/dL
  Treatment Period 1 | -34.81 (34.87) | -39.56 (39.79)
  Treatment Period 2 | -31.27 (33.27) | -41.74 (34.14)

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Levels
Description: Fasting plasma glucose levels were determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 and treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
mg/dL
  Treatment Period 1 | -32.04 (33.95) | -34.48 (32.94)
  Treatment Period 2 | -27.69 (32.19) | -45.51 (35.26)

6. Secondary Outcome: Change From Baseline in 2-hour Post-prandial Glucose (PPG) Levels
Description: 2-hour post-prandial glucose levels were determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 and treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
mg/dL
  Treatment Period 1 | -47.03 (45.85) | -43.36 (48.00)
  Treatment Period 2 | -41.12 (44.77) | -44.03 (43.80)

7. Secondary Outcome: Percent Change From Baseline in Time During 24 Hours With Glucose 70 to 139 mg/dL
Description: Percent change from baseline in time during 24 hours with glucose levels 70 to 139 mg/dL was determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 and treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: PP analysis set included all intent-to-treat participants without a major protocol violation, where ITT population included all participants who received at least one dose of medication and in whom CGM recordings at baseline and after each active treatment were successful.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Percent Change
  Treatment Period 1 | 0.157 (0.134) | 0.191 (0.224)
  Treatment Period 2 | 0.192 (0.214) | 0.182 (0.209)

8. Secondary Outcome: Percent Change From Baseline in Time During 24 Hours With Glucose Greater Than (>) 140 mg/dL
Description: Percent change from baseline in time during 24 hours within the glucose levels >140 mg/dL was determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 and treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Percent Change
  Treatment Period 1 | -0.161 (0.145) | -0.216 (0.257)
  Treatment Period 2 | -214 (0.237) | -0.221 (0.210)

9. Secondary Outcome: Percent Change From Baseline in Time During 24 Hours With Glucose Level > 180 mg/dL
Description: Percent change from baseline in time during 24 hours within the glucose levels >180 mg/dL was determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Percent Change
  Treatment Period 1 | -0.235 (0.204) | -0.212 (0.286)
  Treatment Period 2 | -0.246 (0.232) | -0.251 (0.249)

10. Secondary Outcome: Percent Change From Baseline in Time During 24 Hours With Glucose Level Less Than (<) 70 mg/dL
Description: Percent change from baseline in time during 24 hours within the glucose levels < 70 mg/dL was determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 and treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Percent Change
  Treatment Period 1 | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL. | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL.
  Treatment Period 2 | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL. | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL.

11. Secondary Outcome: Change From Baseline in Time Spent With Glucose Level 70 to 139 mg/dL
Description: Time spent with the glucose level 70 to 139 mg/dL was determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 and treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Minutes
  Treatment Period 1 | 226.64 (193.01) | 275.64 (323.39)
  Treatment Period 2 | 277.00 (309.46) | 261.57 (301.75)

12. Secondary Outcome: Change From Baseline in Time Spent With Glucose Level > 140 mg/dL
Description: Time spent with the glucose level > 140 mg/dL was determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 and treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Minutes
  Treatment Period 1 | -231.98 (208.27) | -310.41 (370.20)
  Treatment Period 2 | -308.68 (341.00) | 318.23 (303.02)

13. Secondary Outcome: Change From Baseline in Time Spent With Glucose Level > 180 mg/dL
Description: Time spent with the glucose level > 180 mg/dL was determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Minutes
  Treatment Period 1 | -338.36 (293.40) | -305.69 (412.30)
  Treatment Period 2 | -354.63 (333.52) | -361.65 (358.27)

14. Secondary Outcome: Change From Baseline in Time Spent With Glucose Level < 70 mg/dL
Description: Time spent with the glucose level < 70 mg/dL was determined over a 6-day period (in order to obtain a continuous 72-hour reading) at baseline and at the end of each active treatment. The participants were analyzed according to treatment received in treatment period 1 and treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Minutes
  Treatment Period 1 | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL. | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL.
  Treatment Period 2 | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL. | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL.

15. Secondary Outcome: Change From Baseline in Percentage of 2 Consecutive Glucose Readings With < 70 mg/dL
Description: The percentage of 2 consecutive glucose readings with < 70 mg/dL were reported. The participants were analyzed according to treatment received in treatment period 1 and treatment period 2 as per the sequence reported in this outcome measure.
Time Frame: Baseline up to End of Treatment Period 1 (Days 22 to 27) and End of Treatment Period 2 (Days 66 to 71)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of readings
Arm/Group | Treatment Sequence AB | Treatment Sequence BA
Number analyzed (Participants) | 31 | 32
Percentage of readings
  Treatment Period 1 | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL. | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL.
  Treatment Period 2 | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL. | NA (NA) — Here, NA signifies that data could not be calculated since there were <5 cases with valid observations of glycemic readings <70 mg/dL.

ADVERSE EVENTS:
Time Frame: Up to 96 Days
Description: Adverse events (AEs) reported are when they occurred under the actual treatment group they were receiving at the AE and not by the randomized sequence. Safety population included all randomized participants who received at least 1 dose of study agent.
Groups:
- Canagliflozin 300 mg: Participants received metformin monotherapy at stable doses (greater than or equal to [>=] 1500 milligram per day [mg/day]) orally once daily with canagliflozin 300 milligram (mg) tablet orally once daily (Treatment A) under fasted condition.
- Sitagliptin 100 mg: Participants received metformin monotherapy at stable doses >= 1500 milligram mg/day orally once daily with sitagliptin 100 mg tablet orally once daily (Treatment B) under fasted condition.
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 7/63 | 2/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin 300 mg (N=63) | Sitagliptin 100 mg (N=63)
Tachycardia (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The main limitation of the study was the sample size limited to demonstrate any significant difference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT03267576/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT03267576/SAP_001.pdf